CLINICAL TRIAL: NCT04085419
Title: Management of Osteoporosis in Patients With Primary Hyperparathyroidism
Brief Title: Osteoporosis in Primary Hyperparathyroidism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Tomaz Kocjan, Professor Tomaz Kocjan, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11111
Record Dates: First submitted 2019-09-02; First posted 2019-09-11 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Primary Hyperparathyroidism; Osteoporosis
Keywords: zoledronic acid; denosumab; primary hyperparathyroidism; osteoporosis
MeSH Terms: conditions — Hyperparathyroidism, Primary; Osteoporosis | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- denosumab (Active Comparator): denosumab 60 mg subcutaneously every 6 months
  Interventions: Drug: Denosumab 60 MG/ML Prefilled Syringe [Prolia]
- zoledronic acid (Active Comparator): zoledronic acid 5 mg intravenously once a year
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Denosumab 60 MG/ML Prefilled Syringe [Prolia] — denosumab 60 mg subcutaneously every 6 months
  Other Names: Xgeva
  Arms: denosumab
Drug: Zoledronic Acid — zoledronic acid 5 mg intravenously once a year
  Other Names: Aclasta
  Arms: zoledronic acid

SUMMARY:
Investigators will prospectively include 40 postmenopausal women with secondary osteoporosis due to primary hyperparathyroidism who have refused surgery. Participants will be randomized in two groups and treated either with zoledronic acid 5 mg iv once a year or with denosumab 60 mg sc every 6 months. Investigators will compare the effect of both drugs on bone turnover markers and basic laboratory parameters after 3, 12 and 24 months of treatment, and on the bone mineral density after 12 and 24 months of treatment. All participants will take cholecalciferol 800 - 1000 IU daily.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (>12 months after last menstrual period) with primary hyperparathyroidism and with osteoporosis on Dual Energy Xray Absorptiometry (DXA) (according to International Society for Clinical Densitometry (ISCD) - criteria) and/or osteoporotic fracture of the vertebra or hip

Exclusion Criteria:

* The patient is not able to give informed consent
* other classic complications of primary hyperparathyroidism (e.g. kidney stones, renal insufficiency)
* serum albumin-corrected calcium level > 2.85 mmol/L (except when the patient is reluctant to undergo surgical treatment)
* osteoporosis treatment less than a year ago, less than two years ago in the case of oral bisphosphonate, less than three years ago in the case of parenteral bisphosphonate
* bilateral hip endoprosthesis
* additional causes for secondary osteoporosis (other than vitamin D deficiency) and pathological laboratory findings that are incompatible with the Summary of Product Characteristics (SmPC) of both medicines
* cancer, except if in stable remission of more than 5 years

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 40 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density after one year of treatment | one year
  Dual-energy X-ray absorptiometry (DXA)
CTX after 3 months of treatment | 3 months
  Unit of Measure: pmol/L
Corrected calcium after 3 months of treatment | 3 months
  Unit of Measure: mmol/L
Bone mineral density after two years of treatment | two years
  Dual-energy X-ray absorptiometry (DXA)
CTX after 12 months of treatment | one year
  Unit of Measure: pmol/L
CTX after 24 months of treatment | two years
  Unit of Measure: pmol/L
PINP after 3 months of treatment | 3 months
  Unit of Measure: µg/L
PINP after 12 months of treatment | one year
  Unit of Measure: µg/L
PINP after 24 months of treatment | two years
  Unit of Measure: µg/L
Bone-specific alkaline phosphatase (BAP) after 3 months of treatment | 3 months
  Unit of Measure: µg/L
Bone-specific alkaline phosphatase (BAP) after 12 months of treatment | one year
  Unit of Measure: µg/L
Bone-specific alkaline phosphatase (BAP) after 24 months of treatment | two years
  Unit of Measure: µg/L
Corrected calcium after 12 months of treatment | one year
  Unit of Measure: mmol/L
Corrected calcium after 24 months of treatment | two years
  Unit of Measure: mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Tomaz Kocjan, MD, PhD, Principal Investigator — UMC Ljubljana
Locations (1):
- Endocrinology Department, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Bone mineral density, bone turnover markers and basic laboratory results will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available in 3 years. They will be available for 5 years.